CLINICAL TRIAL: NCT05667662
Title: Study to Evaluate the Effect of Dose and Duration of Treatment of Itraconazole Administered as a Dry Powder for Inhalation (PUR1900) on Safety, Tolerability, and Potential Outcomes in Adult Patients With ABPA
Brief Title: Study to Evaluate Itraconazole Administered as Inhaled Dry Powder in Adults With Asthma and ABPA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 601-0018
Record Dates: First submitted 2022-12-01; First posted 2022-12-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: ABPA
Keywords: Asthma; Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Asthma; Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PUR1900 40 mg (Experimental): 4 PUR1900 (10 mg itraconazole) Capsules with 20 mg total powder (10 mg itraconazole plus 10 mg excipients) administered via oral inhalation, using the RS01 Monodose inhaler once daily for 112 days at approximately the same time each day.
  Interventions: Drug: Itraconazole Powder
- PUR1900 20 mg (Experimental): 2 PUR1900 (10 mg itraconazole) Capsules with 20 mg total powder (10 mg itraconazole plus 10 mg excipients) and 2 Placebo Capsules with with 11.8 mg total powder (excipients only) administered via oral inhalation, using the RS01 Monodose inhaler once daily for 112 days at approximately the same time each day.
  Interventions: Drug: Itraconazole Powder
- Placebo (Placebo Comparator): 4 Placebo Capsules with with 11.8 mg total powder (excipients only) administered via oral inhalation, using the RS01 Monodose inhaler once daily for 112 days at approximately the same time each day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itraconazole Powder — Capsules with 20 mg total powder (10 mg itraconazole plus 10 mg excipients)
  Other Names: PUR1900
  Arms: PUR1900 20 mg; PUR1900 40 mg
Drug: Placebo — Capsules with 11.8 mg total powder (excipients only)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about PUR1900 as an inhaled, antifungal therapeutic for the treatment of allergic bronchopulmonary aspergillosis (ABPA) in patients with asthma. The main questions it aims to answer are:

1. Is PUR1900 safe and well tolerated in adults with asthma and ABPA?
2. Is there an effect of daily administration of PUR1900 on potential outcome measures in adults with asthma and ABPA?
3. Is there fungal resistance to A. fumigatus?

This study includes a 28-day screening period, a 112-day (16-week) treatment period, and a 56-day (8 week) observation period.

Participants will take either 40mg of PUR1900, 20 mg of PUR1900 or Placebo for 112 days and complete an eDairy, answer questions about their asthma and complete peak respiratory flow measurements at home. They will come to the clinic approximate once a month during the treatment period and complete study assessments. At the end of the observation period participants will complete one more clinic visit. Participants who complete this study may be given the opportunity to continue on study drug in an open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female, ≥18 years old at the time of signing the informed consent.
* BMI of ≥18.0 and <40.0 kg/m2 at screening.
* Has a diagnosis of asthma, as per the Global Initiative for Asthma (GINA) 2018 update
* Has a confirmed diagnosis of ABPA, based on the modified International Society for human and Animal Mycology (ISHAM) ABPA working group 2013 and 2021 criteria including a history of or documentation at screening of serum IgE ≥ 500 IU/mL and A. fumigatus-specific IgE>0.35KUA/L, or above normal IgE antibody to A. fumigatus, or a positive immediate skin test and at least 2 of the 3 following supportive criteria: eosinophil count >500 cells/µL; A. fumigatus-specific IgG >27 mgA/L or presence of precipitating (or above normal immunoglobulin G [IgG]) antibody to A. fumigatus; consistent radiographic opacities or bronchiectasis on chest CT.
* Is currently considered to be in one of the following stages of ABPA: Stage 2 (Response), Stage 4 (Remission), Stage 5a (Treatment-dependent ABPA), or Stage 5b (Glucocorticoid-dependent asthma).
* At least 1 exacerbation requiring a systemic glucocorticosteroid(s) in the 12 months prior to Screening. For patients on a biologic agent, at least one exacerbation requiring a systemic glucocorticosteroid(s) must have occurred at least 3 months after the initiation of the biologic agent.
* Has a serum IgE ≥500 IU/mL at screening.
* Has a documented stable asthma medication regimen during the 28 days prior to the first dose of study drug ; applicable asthma medications can include but are not limited to the following: inhaled short-acting beta agonist (SABA), inhaled long-acting beta agonist (LABA), and leukotriene receptor antagonist (LTRA) use and inhaled and/or oral glucocorticosteroids. SABA use during this period should be mostly within a stable range (e.g., 2 puffs 2 to 4 times a day) and should not exceed 8 puffs a day on 2 out of 3 consecutive days.
* Can perform a valid, reproducible spirometry test with demonstration of a prebronchodilator FEV1 ≥50% of predicted normal for age, sex, race, and height at a screening visit.
* Can demonstrate the correct inhalation technique and achieve a minimum inspiratory flow rate of 45 L/min for the use of the delivery device at screening and before dosing on Day 1.
* Is willing and able to comply with all study procedures and assessments, including scheduled visits, drug dosing plan, study procedures, laboratory tests, and study restrictions.
* Subjects who are sexually active, male subjects able to father a child, and female subjects of childbearing potential must agree to follow contraception requirements.

Exclusion Criteria:

* Currently requiring medications that are sensitive substrates for CYP3A4-mediated metabolism or medications that are contraindicated with oral itraconazole.
* Has evidence of ventricular dysfunction, such as congestive cardiac failure (New York Heart Association functional class III or IV), or a history of congestive cardiac failure. N-terminal pro B-type natriuretic peptide (NT pro BNP) will be checked at screening only. A subject with a confirmed value of >400 pg/mL will not be eligible to participate.
* Has used any systemic azole antifungal agent in the 6 weeks before first dose of study drug.
* Has discontinued previously administered biologic agent(s) in the 3 months prior to screening.
* Has a history of life-threatening asthma within the last 24 months, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, and/or hypoxic seizures.
* Has a current diagnosis of any chronic airway disease other than asthma, ABPA, or bronchiectasis believed to be related to ABPA, such as chronic obstructive pulmonary disease, pulmonary fibrosis, cystic fibrosis, or Churg-Strauss syndrome. A subject whose predominating clinical disease burden is related to bronchiectasis (e.g., a subject with 2 or more infective exacerbations of bronchiectasis in the past 12 months or a subject with chronic colonization with Pseudomonas aeruginosa) will be excluded. Refer to Appendix 4 for definition of bronchiectasis exacerbations.
* Had an occurrence of clinically significant bacterial, viral, or fungal infection that required systemic (oral or intravenous) antibiotics, antivirals, or antifungals within the 28 days before screening. Topical treatments, other than antifungals, are allowed.
* Had an occurrence of asthma or ABPA exacerbations within the 28 days before screening.
* Has the presence of hoarseness or oropharyngeal candidiasis at screening.
* Had a major trauma or surgery within the last 28-days before screening.
* Has a history of any clinically significant cardiovascular, renal, hepatic, or gastrointestinal disease or neurological or psychiatric disorder endocrine, immunological, or autoimmune disease or other medical condition that would affect the subject's safety or confound the assessment of study endpoints as judged by the Investigator.
* Has a history of any clinically significant drug or alcohol abuse in the past 6 months before screening, as judged by the Investigator.
* Has current inhaled tobacco/nicotine or inhaled marijuana use or history of smoking or vaping including tobacco or marijuana within the last 6 months before screening.
* Has a history of any clinically significant drug or alcohol abuse in the past 6 months before screening, as judged by the Investigator.
* Has current tobacco or inhaled marijuana use or history of smoking or vaping including tobacco or marijuana within the last 6 months before screening.
* Has a history of allergic or hypersensitivity reaction or serious adverse reaction after dosing of itraconazole or other antifungal azoles.
* Has a history of serious adverse reaction or known serious hypersensitivity to any of the formulation excipients.
* Has a positive urine test result for drugs of abuse or cotinine at screening (unless, in the opinion of the Investigator, this can be explained by the subject's current medications). Note that results that are positive for a drug of abuse or cotinine may be acceptable for drugs that have been obtained by legal means or non-inhaled tobacco/nicotine product use.
* At screening, has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x upper limit of normal (ULN), white blood cell (WBC) count > 20,000 X 109/L, absolute neutrophil count <1000 cells/L, platelet counts <100,000 to or >500,000 X 109/L, or hemoglobin <10 g/dL
* Is a female of childbearing potential who is pregnant or lactating or who plans to become pregnant during the study. All female subjects must have a negative pregnancy test at screening and pre dose on Day 1. A woman is of childbearing potential unless she is either permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, bilateral tubal occlusion/ligation, endometrial ablation) or postmenopausal (had no menses for 12 months without an alternative medical cause).
* Has a 12-lead ECG demonstrating a mean QT interval corrected by the Fridericia formula (QTcF) >450 msec for a male subject or >470 msec for a female subject at screening. A repeat triplicate ECG is allowed if a mean QTcF >450 msec for males and >470 msec for females is recorded at Visit 1.
* Has a planned or elective surgery, hospitalizations, or participation in other interventional studies any time during the study that may interfere with study logistics or safety.
* Has donated or had a loss of greater than 400 mL of blood within the 3 months before screening.
* Has other social, psychiatric, surgical, or medical conditions or screening laboratory abnormalities that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the Investigator, would make the subject inappropriate for entry into the study.
* Received any investigational medical product in a clinical research study within the previous 3 months before first dose of study drug.
* Is a study site employee, an immediate family member of a study site employee, or a Sponsor employee.
* Has previously received PUR1900.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 168 days
  Review of TEAEs from time of consent to study completion.
Safety spirometry assessments | 168 days
  FEV1 (the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration), FVC (liters), and PEFR (L/min) measurements compared to baseline.
Vital sign measurements | 168 days
  Vital signs measurements collected before exposure, during and after treatment and compared to baseline. Vital sign measurements will include respiratory rate (bpm), blood pressure (mmHg), heart rate (bpm), oxygen saturation (by pulse oximetry), and oral or tympanic temperature (°C).
Physical examinations | 168 Days
  At screening, a complete physical examination will be performed which includes measurement of height (cm), weight (kg) and evaluation of appearance; skin; head and neck; eyes, ears, nose, and throat; chest and lungs; heart; abdomen; neurological system; and extremities.
Clinical safety laboratory test results | 168 days
  Hematology, serum chemistry, or urinalysis test results (normal, abnormal, clinical significance) compared to baseline.
Cardiac safety monitoring | 168 days
  Electrocardiogram (ECG) recordings collected before exposure, during and after treatment. Electrocardiogram measurements will include heart rate and PR, RR, QRS, and QT intervals, as well as the QTcF and compared to baseline.

SECONDARY OUTCOMES:
Magnitude of effect of daily administration of PUR1900 - Spirometry | 168 days
  Changes in measured Forced Expiratory Volume (FEV1) over time compared to baseline
Magnitude of effect of daily administration of PUR1900 - Patient Reported Outcomes (ACQ) | 168 days
  Responses to the Asthma Control Questionnaire (ACQ) sored from 0-6 with 0 being totally controlled and 6 being extremely poorly controlled compared to baseline.
Magnitude of effect of daily administration of PUR1900 - Patient Reported Outcomes (AQLQ(s) 12+) | 168 days
  Responses to the Asthma Quality of Life Questionnaire with scores ranging 1-7 and higher scores indicating better quality of life compared to baseline.
Frequency of asthma exacerbations versus baseline | 168 days
  Occurrence of asthma exacerbations before, during, and after treatment with PUR1900

OTHER OUTCOMES:
Fungal resistance to Aspergillus fumigatus | 168 days
  Fungal susceptibility of sputum samples collected at the before and after anti-fungal treatment to determine resistance risks using the EUCAST microdilution method

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cabell, MD, Study Director — Pulmatrix Inc.
Locations (18):
- United States (8):
  - University of Alabama Medical Center at Birmingham, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - Jonathan Corren, MD, Santa Monica, California
  - Bensch Clinical Research, Stockton, California
  - Southern Illinois University Center for Clinical Research, Springfield, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Baylor University Medical Center, Dallas, Texas
  - UTMB Health, Galveston, Texas
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Mater Hospital Brisbane, Respiratory Research Group, South Brisbane, Queensland
  - Royal Perth Hospital, Perth, Western Australia
- France (3):
  - CHU Pontchaillou, Rennes, Cedex 9
  - Nouvel Hôpital Civil, Strasbourg, Strasbourg Cedex
  - CHU de Marseille Hôpital Nord, Marseille
- United Kingdom (4):
  - University Hospitals Birmingham - Heartlands Hospital, Birmingham, West Midlands
  - CPS Research Limited, Glasgow
  - Royal Brompton Hospital, London
  - University Hospital of South Manchester - Wythenshawe Hospital,, Manchester